CLINICAL TRIAL: NCT03788278
Title: An Advanced Digital Phenotype System Among People Suffering From Post-traumatic Stress Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nadav Goldental (Other)
Responsible Party: Sponsor-Investigator, Nadav Goldental, Principal investigator, The Chaim Sheba Medical Center
Organization: The Chaim Sheba Medical Center (Other)
Other Study IDs: SHEBA-5184-18-SMC
Record Dates: First submitted 2018-12-03; First posted 2018-12-27 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Digital psychiatry
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTSD patients: Participants will attend clinical surveillance once every week or two. During the follow-up period, the participant will be checked as usual and will have to fill in questionnaires.
  Participants will be required to wear the smart watch at all times and will need to recharge it at least once every three days.
  Participants will be required to answer digital questionnaires twice a day via smartphone.
  Interventions: Device: BioBeat
- Non PTSD participants: Participants will attend clinical surveillance once every week or two. During the follow-up period, the participant will be checked as usual and will have to fill in questionnaires.
  Participants will be required to wear the smart watch at all times and will need to recharge it at least once every three days.
  Participants will be required to answer digital questionnaires twice a day via smartphone.
  Interventions: Device: BioBeat

INTERVENTIONS:
Device: BioBeat — The watch incorporates sensors, a battery, a software system, memory components, and a communications component. the watch will be worn 24 hours a day, 7 days a week.

SUMMARY:
Psychiatric diagnosis is based mainly on questioning the patient and subjective impression rather than a quantitative assessment. The assessment is usually done with long time intervals between assessments and arbitrary in relation to the clinical course of the disorder. Post-traumatic stress disorder has physiological, physical, and behavioral manifestations. These changes appear as a response to different situations during the day and can be measured directly and indirectly in order to obtain an objective, quantitative and fuller picture of the severity and changes in the disorder. This is a non-interventional pilot study, using a system that collects data through wearable sensors and smartphone over a long period of time for patients suffering from PTSD and enables data analysis and characterization of a personal digital phenotype using a dedicated algorithm. Based on this pattern, the investigators will attempt to support the establishment of the PTSD diagnosis. During the course of the study, the therapeutic procedure will not be affected by the study and will be independent of the research.

ELIGIBILITY:
Inclusion Criteria for study group:

* Current PTSD diagnosis based on DSM-5. We will aim to recruit patients with Clinically Administered PTSD Scale (CAPS)- 5, medium severity and up.
* A person who is being monitored by the Ministry of Defense PTSD clinic at the Sheba Medical Center.
* Proper ability to give informed consent.
* A person with a smartphone that is not hacked with an Android version 2.3 or higher (relevant to smartphones manufactured since 2011).

Inclusion Criteria for control group:

* Proper ability to give informed consent.
* A person with a smartphone that is not hacked with an Android version 2.3 or higher (relevant to smartphones manufactured since 2011).

Exclusion Criteria for study group:

* A person defined as a violent or suicidal person (significant events of physical violence or suicidal behavior in the past year, according to the treating psychiatrist professional opinion).
* An active or terminal oncology disease or a dialysis patient.
* A person who is not independent or reports that he/she will not meet the requirement to wear the watch, recharge it or any other requirement arising from the use of the watch.
* A person without a smartphone that is not hacked or without Android version 2.3 or higher (relevant to smartphones manufactured since 2011).

Exclusion Criteria for control group:

* Current mental health diagnosis.
* A person defined as a violent or suicidal person (significant events of physical violence or suicidal behavior in the past year, according to the treating psychiatrist professional opinion).
* An active or terminal oncology disease or a dialysis patient.
* A person who is not independent or reports that he/she will not meet the requirement to wear the watch, recharge it or any other requirement arising from the use of the watch.
* A person without a smartphone that is not hacked or without Android version 2.3 or higher (relevant to smartphones manufactured since 2011).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years and older from both sexes. The study group will include 25 participants with a diagnosis of PTSD. The participants will be recruited from among the patients at the Ministry of Defense clinic at the Sheba Medical Center. The control group will consist of 25 participants recruited from medical staff and students from the Sheba Medical Center and Tel-Aviv University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-20 (Estimated); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlations between data changes and PTSD clinical symptoms | Three months
  Investigators will use a wearable smart watch to collect physiological data (Heart Rate, Cardiac Output, Blood Pressure, Respiratory Rate, Steps Counter, Electro-Dermal Activity) and will use psychiatric rating score (CAPS 5, CGI, PHQ-SADS) to determine changes in clinical symptoms. The investigators will look for correlations between the collected physiological data and the clinical symptoms according to the psychiatric rating scales

IPD SHARING:
Plan to Share IPD: No